CLINICAL TRIAL: NCT00630630
Title: A Multicenter, Double-blind, Placebo-controlled, Parallel Group Study of the Safety and Efficacy of Levetiracetam in the Adjunctive Treatment of Adult Female Subjects (18 to 40 Years of Age) With C1 Catamenial Epilepsy
Brief Title: Study on Safety and Efficacy of Levetiracetam in the Adjunctive Treatment of Female Subjects With C1 Catamenial Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01088
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Levetiracetam
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levetiracetam
  Other Names: Keppra, ucbL059
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
The relationship between hormone cycling/fluctuations and the occurrence of seizures in women has received considerable discussion in the medical literature. This study investigated the efficacy and tolerability of LEV treatment for subjects with catamenial exacerbation of partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-nursing females between the ages of 18 - 45 years of age;
* out-patients with epilepsy experiencing uncontrolled simple and/or complex partial seizures with or without secondary generalization for a minimum of 2 years;
* classifiable epilepsy according to the International Classification of Epileptic Seizures;
* minimum of 2 seizures per 4 weeks during the Baseline Period, without exceeding 100 seizures per 4 weeks. The majority of seizures (>50%) must be partial onset, with or without secondary generalization;
* exhibited, during the Baseline Period, a catamenial epilepsy type C1 pattern defined as at least a 70% increase of weekly seizure frequency during the menstrual phase compared to the luteal and follicular phases combined;
* concurrent C2 catamenial epilepsy, defined as a 70% increase in daily seizure average during the ovulatory phase in comparison to the follicular and luteal phases combined, was permitted;
* taking a minimum of one and a maximum of two antiepileptic drugs at a stable dose for a period of 4 weeks prior to the selection visit and during the duration of the trial;
* vagal nerve stimulator (VNS) was permitted.

Exclusion Criteria:

* using felbatol and presented clinically significant abnormalities with WBCs, RBCs, platelets, and/or hepatic function during felbatol treatment, and taking felbatol less than one year from the date of the Selection Visit;
* partial onset seizures uncountable due to clustering during the last 3 months;
* hormonal contraceptives that block menses within 6 months of the selection visit with no washout period permitted;
* menstrual cycle length less than 21 days and greater than 35 days during the baseline evaluation;
* alternative medications documented or purported to impact reproductive hormone levels, within the prior 2 months with no washout period permitted;
* significantly irregular menstrual cycles or a history of frequent amenorrhea defined as two episodes within the preceding 6 months;
* not taking hormonal contraceptives with more than one anovulatory cycle during the Baseline Period;
* clinically significant medical condition requiring treatment, except for the study indication, which would prevent clear interpretation of the study results;
* using the following classes of medications influencing the central nervous system: antipsychotics (typical and atypical), psychostimulants (except those containing methylphenidate, dextroamphetamine, or amphetamine used in the treatment of Attention Deficit Disorder), and hypnotics;
* chronically dosing with benzodiazepines;
* hospitalized for depression within 3 months prior to the selection visit.
* history of attempting suicide within the last 3 years, or suicidal ideation within the last 3 months;
* recent history (within the past two years) or presence of significant alcohol abuse or drug abuse;
* clinical history of significantly impaired renal function with a estimate of creatinine clearance below 80 ml/min;
* history of clinically significant cardiac conditions;
* ALT/SGPT, AST/SGOT, alkaline phosphatase, or ?-GT value of more than 3 times the upper limit of the central laboratory reference value;
* presence of a terminal illness;
* presence of any clinically significant allergic condition to levetiracetam or pyrrolidone derivatives;
* neutrophil count of less than 1800 per ?L.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2002-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Percent change in catamenial seizure frequency.

SECONDARY OUTCOMES:
Responder rate
Number of days free from seizures per week
Ratio of catamenial seizure frequency to non-catamenial seizure frequency
Catamenial seizure frequency during each cycle
Seizure frequency of catamenial and non-catamenial combined
Non-catamenial seizure frequency
Catamenial seizure frequency separately for ovulatory and anovulatory cycles
Safety

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)